CLINICAL TRIAL: NCT03691597
Title: Patient Satisfaction ,Marginal Integrity ,Shade Matching and Gingival Health of Zirconia Reinforced Lithium Silicate Bridges Cemented Using Bioactive Cement and Adhesive Resin Cement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nihal anwar Mohamed haffour, Assistant lecturer ,fixed prosthodontics department,faculty of oral and dental medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-09-41
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Patient Satisfaction ,Marginal Integrity, Shade Match and Gingival Health

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adhesive resin cement (Active Comparator): type of cement used for cementation of crowns have a good adhesion bond
  Interventions: Diagnostic Test: improved patient satisfaction ,marginal integrity, shade match and gingival health
- Bioactive cement (Experimental): recent cement improve the marginal integrity
  Interventions: Diagnostic Test: improved patient satisfaction ,marginal integrity, shade match and gingival health

INTERVENTIONS:
Diagnostic Test: improved patient satisfaction ,marginal integrity, shade match and gingival health — For both groups N.Awill make a recall visit after6 months and after 12 months:
  1. Patient satisfaction will be performed according to questionnaire after One year.Questionnaire will contain several questions that evaluate patient satisfaction.
  2. The color will be measured using spectrophotometer Vita easy shade in the same delivery visit ,after 6months and after one year .
  3. Images will be captured using digital handheld light microscope (Celestron 5 Megapixel Resolution, USA) that is fixed on a film holder on a specific distance for the standardization of all the images will be captured by the microscope for all the patients.(22)
  4. Images will be analyzed using imageJ software to measure marginal gap.
  5. Gingival health will be measured using G

SUMMARY:
Bioactive cement have been introduced recently into the market according to the manufacture it is assumed that it stimulates mineral apatite formation and the natural remineralization process at the material-tooth interface that knits together the restoration and the tooth, penetrates and fills micro-gaps, reduces sensitivity, guards against secondary caries, and seals margins against microleakage

DETAILED DESCRIPTION:
To evaluate the cement type (bioactive cement and adhesive resin cement ) on Patient satisfaction ,marginal integrity ,shade matching and gingival health of cemented zirconia reinforced lithium silicate restoration .

PICOTS:

P: patients with missing anterior teeth that needs fixed restoration . I: Bioactive cement. C: adhesive resin cement. O: patient satisfaction ,margin integrity ,shade matching and gingival health T: 1 year

ELIGIBILITY:
Inclusion Criteria:" Permanent anterior teeth. " Vital teeth with Absence of clinical diagnosis of pulp exposure, periapical pathosis, fistula, swelling of periodontal tissues, abnormal tooth mobility, and history of spontaneous pain or sensitivity to pressure.

" Healthy appearance of adjacent gingiva.

-

Exclusion Criteria:

* Periapical pathosis, Signs of pulpal pathology, Severe periodontal affection these cases are not indicated for full coverage restoration.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
margin integrity | one year
  accuracy of adaptation of restoration and close marginal gap

CONTACTS AND LOCATIONS:
Overall Officials: Gihan GN elnagar, professor, Study Director — faculty of oral and dental medicine Cairo university

IPD SHARING:
Plan to Share IPD: No
Bioactive cement have been introduced recently into the market according to the manufacture it is assumed that it stimulates mineral apatite formation and the natural remineralization process at the material-tooth interface that knits together the restoration and the tooth, penetrates and fills micro-gaps, reduces sensitivity, guards against secondary caries, and seals margins against microleakage